CLINICAL TRIAL: NCT02876016
Title: Cerebral Bases Bodily Representations: Imaging Approach by Functional Magnetic Resonance, Cortical Stimulation Corticographie and Surgery Awake
Brief Title: Cerebral Bases Bodily Representations
Acronym: EBA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-34; 2014-A01449-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Glial Tumors
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- awake brain surgery (Experimental): Exploration of the cortical area of the brain awake surgery
  Interventions: Device: functional MRI

INTERVENTIONS:
Device: functional MRI — locate the cerebral bases in functional imaging

SUMMARY:
Bring elements of understanding to the study of brain organization bodily representations. The body is organized into multiple, distinct levels of representation. The body schema is an unconscious and dynamic representation of his body, updated constantly, resulting from the convergence of multiple sensory information, which articulates with the motor systems to participate in the genesis of the action. The self-image corresponds to a more abstract representation of the body, covering symbolic and imaginary aspects drawn from the emotional life of the individual. Finally, the body of another person engages simultaneously shared and differential representational systems that allow understanding the actions of others while preserving the identity of the agent responsible for the action. These various bodies represented subtly interacting and participating in equilibrium, the self-awareness building as being curious, social and acting. Brain organization bodily representations remains a fundamental question still poorly explored that is of major scientific interest because of its influence on identity and social construction, and the serious repercussions that are their problems, also for the individual and society. This project aims to deepen this hypothesis using a methodology combining functional imaging and awake surgery. The richness of this project lies in the innovative methods of investigation, and in the plurality of disciplines (neuropsychology, neurophysiology, neuroimaging and neurosurgery) and teams (clinical and research) grouped for wear.

The subjects enrolled in this study are all candidates in patients with awakened provided surgery for therapeutic reasons, and volunteer to participate in this experiment. Awake neurosurgery is for patients with glial tumors, but also brain metastases and intra-parenchymal cavernomas. A first experimental session will be held in pre-operative period. Patients realize a functional magnetic resonance imaging (fMRI) brain to define a precise functional mapping of cortical structures, including lateral occipital, involved in body representation. The second experimental session will be conducted in the neurosurgical intervention, practiced one to four weeks later.

This dual approach that combines the functional stimulation of a cortical area (imaging) and functional inhibition (in surgery) allows you to make extremely robust scientific arguments about the causal relationships linking structure and function

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Candidate awake in a long surgery
* Carrying on an original tumor glial parietal or temporal
* Normal global cognitive efficiency score greater than or equal to 27

Exclusion Criteria:

* Patient ambidextrous or left
* Non glial tumor
* Tumor not involving the temporal or parietal lobes
* Consumption of non-drug substance
* Visual perceptual disorder and or space
* Global Cognitive Impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
localization of cortical areas | 36 months
  Detection the activity of neurons by the signal of functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Olivier FELICIAN, PU-PH, Principal Investigator — Assitance Publique Hôpitaux de Marseille
Locations (1):
- Assitance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No